CLINICAL TRIAL: NCT07402239
Title: The Study of a tHerApeutic and monitoRing Device iMplanted at the Atrial Septum prOvides Heart Failure maNagement in sYmptomatic Patients (HARMONY Trial)
Brief Title: HARMONY Trial : To Evaluate a Therapeutic and Monitoring Device(NOVAtria System) for Heart Failure Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: United Innomed(Shanghai) Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHF101-004A
Record Dates: First submitted 2026-01-29; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment (Experimental): Treatment arm patients will undergo a right heart catheterization and invasive echocardiography to determine study eligibility and TEE guided trans-septal puncture and NOVAtria® system procedure
  Interventions: Device: NOVAtria System
- Control (Other): Control arm patients will undergo a diagnostic right heart catheterization and invasive echocardiography to determine study eligibility, but will not have transseptal catheterization or device implantation
  Interventions: Other: Control
- Roll in (Experimental): Roll in arm patients will undergo a diagnostic right heart catheterization and invasive echocardiography to determine study eligibility followed by transseptal catheterization and NOVAtria® system procedure
  Interventions: Device: NOVAtria System

INTERVENTIONS:
Device: NOVAtria System — The NOVAtria System, therapeutic and monitoring device will be implanted at interatrial septum with minimally invasive cardiac catheterization procedure
  Arms: Roll in; Treatment
Other: Control — Right heart catheterization and TEE
  Arms: Control

SUMMARY:
The objective of the HARMONY trial is to evaluate the safety and efficacy of implantable left atrial pressure sensor and interatrial shunt system for the treatment of chronic heart failure with reduced left ventricular ejection fraction (HFrEF, EF ≤ 40%) and New York Heart Association(NYHA) functional Class II or Class III who at baseline are treated with guideline-directed drug and device therapies.

ELIGIBILITY:
Main Inclusion Criteria：

* Age ≥ 18 years old
* Clinically diagnosed with chronic heart failure
* Receiving guideline directed medical and device therapy (GDMT) for heart failure
* Left ventricular ejection fraction (LVEF) ≤ 40% assessed by echocardiography
* New York Heart Association (NYHA) functional class II or III, with NYHA II criteria met simultaneously; for NYHA III, at least one of the following must be satisfied:

  1. At least one hospitalization for heart failure within the past 12 months;
  2. Elevated BNP or NT-proBNP within 3 months prior to enrollment (under normal sinus rhythm, NT-proBNP > 900 pg/mL; under atrial fibrillation, NT-proBNP > 1500 pg/mL; under normal sinus rhythm, BNP > 300 pg/mL; under atrial fibrillation, BNP > 500 pg/mL; BNP not applicable if the patient is using ARNI);
* Able to perform 6-minute walk test (6MWT), with a distance between 100 meters and 450 meters

Main Exclusion Criteria

* Currently in an acute decompensation of chronic heart failure (hospitalization within 2 weeks prior to enrollment), refractory end-stage heart failure, or on the waiting list for heart transplantation (including LVAD indication);
* BMI > 40 kg/m² or < 18.5 kg/m²;
* Systolic blood pressure <90 or ≥160 mmHg
* Moderate or severe aortic or mitral stenosis, or planned during the trial intervention for severe regurgitation of the aortic, mitral, tricuspid, or pulmonary valves;
* Coronary artery disease requiring revascularization;
* Hypertrophic cardiomyopathy, active myocarditis, cardiac tamponade or large pericardial effusion, congenital heart disease, or other causes of heart failure
* History of stroke, transient ischemic attack (TIA), deep vein thrombosis (DVT), or pulmonary emboli within the past 3 months
* Severe chronic lung disease requiring oxygen therapy or long-term corticosteroids;
* Surgery involving atrial septal puncture within 3 months before enrollment (e.g., mitral repair, atrial fibrillation ablation, LAA closure);
* Significant RV dysfunction - TAPSE <12mm or RVFAC ≤25%
* eGFR <25 ml/min/1.73 m^2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Primary Safety endpoint | 30-days after randomization
  Safety-Percentage of Treatment patients experiencing major device-related adverse events.Percentage of Treatment group patients experiencing any device-related Major Adverse Cardiovascular or Neurological Events (MACNE) during the first 30-days after randomization, compared to a pre-specified Performance Goal
Composite Primary Effective endpoint | Follow-up duration at endpoint analysis ranges from a minimum of 12 to a maximum of 24 months
  Effectiveness-Hierarchical composite of death, heart transplant or left ventricular assist device (LVAD) implantation, HF hospitalizations, worsening HF events treated as an outpatient, and change in 6WMT

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medcine, Hangzhou, Zhejiang, China